CLINICAL TRIAL: NCT07142915
Title: A Prospective Randomized Controlled Trial on the Effect of Light-Blocking Lenses on Emmetropization in Hyperopic Children
Brief Title: Effect of Light-Blocking Lenses on Pediatric Hyperopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jingrong Li, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025KYPJ081
Record Dates: First submitted 2025-08-18; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hyperopia
Keywords: hyperopia; light-blocking lenses; emmetropization; visual function
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Subjects will be instructed to wear light-blocking lenses full-time for 12 months. Scheduled follow-up examinations will be conducted at 6 months (±15 days) and 12 months (±15 days) after lens fitting. Replacement of the lenses will be arranged if a refractive change greater than 0.50 diopters is observed, or in cases of severe lens damage.
  Interventions: Other: light-blocking lenses
- Control Group (Placebo Comparator): Subjects will be instructed to wear single-vision lenses full-time for 12 months. Scheduled follow-up examinations will be conducted at 6 months (±15 days) and 12 months (±15 days) after lens fitting. Replacement of the lenses will be arranged if a refractive change greater than 0.50 diopters is observed, or in cases of severe lens damage.
  Interventions: Other: single-vision lenses

INTERVENTIONS:
Other: light-blocking lenses — Subjects will be instructed to wear light-blocking lenses full-time for 12 months.
  Arms: Intervention Group
Other: single-vision lenses — Subjects will be instructed to wear single-vision lenses full-time for 12 months.
  Arms: Control Group

SUMMARY:
This study aims to assess the efficacy of light-blocking lenses in facilitating emmetropization in children with hyperopia and to explore their influence on various aspects of visual function.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 years or older and 12 years or younger;
* Spherical refractive error in both eyes between +3.0 D and +7.5 D, cylindrical refractive error between -2.0 D and 0 D; interocular difference in spherical power less than 1.5 D and in cylindrical power no greater than 1.0 D;
* Best-corrected visual acuity of 0.0 logMAR or better in both eyes;
* Ocular deviation with spectacles less than 10 prism diopters;
* Has been wearing standard single-vision spectacles regularly for more than six months;
* In good general health, capable of receiving the study intervention, and willing to comply with the study protocol;
* Written informed consent obtained from both the parent/guardian and the child, with agreement to comply with all study procedures and maintain follow-up availability throughout the study period;

Exclusion Criteria:

* History of ocular trauma or eye surgery;
* Presence of pathological abnormalities on anterior or posterior segment examination, or a history of organic ocular diseases such as cataract, glaucoma, corneal disease, or fundus disorders;
* Intraocular pressure greater than 21 mmHg;
* Presence of systemic diseases or other conditions deemed unsuitable for study participation;
* Any other condition deemed inappropriate for participation in the clinical trial by the investigator;

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Axial length | At baseline, 6 months, and 12 months
  measured by optical biometer

SECONDARY OUTCOMES:
Refractive error | At baseline, 6 months, and 12 months
  measured by cycloplegic refraction
Best-corrected visual acuity | At baseline, 6 months, and 12 months
  measured by visual acuity chart
Intraocular pressure | At baseline, 6 months, and 12 months
  measured by non-contact tonometer
Angle of deviation | At baseline, 6 months, and 12 months
  measured by alternate cover test with prism
Contrast sensitivity | At baseline, 6 months, and 12 months
  measured by quick contrast sensitivity function test
Stereopsis | At baseline, 6 months, and 12 months
  measured by stereotest booklet
Accommodative function | At baseline, 6 months, and 12 months
  measured by phoropter
Intervention questionnaire | At baseline, 6 months, and 12 months
  measured by questionnaire

OTHER OUTCOMES:
Height | At baseline, 6 months, and 12 months
  measured by ruler
Weight | At baseline, 6 months, and 12 months
  measured by weighing scale
Choroidal thickness (optional) | At baseline, 6 months, and 12 months
  measured by OCT, optional

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No